CLINICAL TRIAL: NCT03940001
Title: A Study of Anti-PD-1 Antibody, Sintilimab Plus Chemoradiation Before Surgery for Esophageal Cancer
Brief Title: A Study of Sintilimab Plus Chemoradiation Before Surgery for Esophageal Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZJCH1903
Record Dates: First submitted 2019-05-04; First posted 2019-05-07 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-05

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — sintilimab; CP protocol; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- arm (Experimental): Biological: Sintilimab For weight <60kg, 3mg/kg IV Q3W day 1, and for weight≥60kg, 200mg IV Q3W day 1
  Drug: Paclitaxel 50 mg/m^2 IV Q3W day 1, day 8 and day 15
  Drug: carboplatin AUC: 2 IV Q3W day 1, day 8 and day 15
  Radiotherapy:
  1.8 Gy/fraction ×23 fractions Monday to Friday total dose of 41.4 Gy
  Interventions: Biological: Sintilimab; Drug: carboplatin/paclitaxel; Radiation: Radiation

INTERVENTIONS:
Biological: Sintilimab — Other Name: (IBI308)
Drug: carboplatin/paclitaxel — carboplatin AUC 2/paclitaxel 50 mg/m2 weekly
Radiation: Radiation — IMRT or VMAT

SUMMARY:
The purpose of this study is to test the the efficacy and safety of sintilimab in combination with chemoradiation before surgery for esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed esophageal squamous carcinoma
* 18≤age≤75
* ECOG PS is 0-1
* TanyN+M0 or T3-4NanyM0 tumors
* Patients must have surgically resectable disease treatable by esophagectomy, as assessed by a thoracic surgeon
* No prior chemotherapy,radiotherapy and immunotherapy
* Disease must be clinically limited to the esophagus
* No esophageal perforation and no active esophageal bleeding
* No interstitial pneumonia or history of interstitial pneumonia
* FEV1>1.2L
* Adequate organ function defined at baseline as: WBC ≥3,000/ L，ANC ≥1,500/ L，Platelets ≥100,000/ L，Hb ≥9 g/dl； Calculated creatinine clearance >40 ml/min using Cockcroft-Gault method: Males: Creatinine CL = Weight (kg) x (140 - Age) . (mL/min) 72 x serum creatinine (mg/dL)Female：Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)；Total serum bilirubin ≤1.5 mg/dL， AST/ALT ≤2.5× upper limit of normal，Mean QT interval corrected for heart rate (QTc) <470 ms calculated from 3 ECGs using Frediricia's Correction
* Able to provide written informed consent
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

* Previous treatment with chemotherapy, radiotherapy or immunotherapy
* Cervical esophageal cancer
* Esophageal perforation or active esophageal bleeding
* Interstitial pneumonia or history of interstitial pneumonia
* Patients with evidence of metastatic disease
* Chronic Hepatitis B or C infection (e.g. Hepatitis B surface Ag positive or detectable viral load for Hepatitis B or C). Patients with prior evidence of Hepatitis B or C without active infection are eligible
* Autoimmune diseases (such as systemic lupus erythematosus, rheumatoid rthritis, inflammatory bowel disease, autoimmune thyroid disease), but allow the following diseases to enter the next stage of screening: type I diabetes, skin diseases without systemic treatment (such as vitiligo, psoriasis)
* 14 days before the first dose, the patient had an active infection that required systemic treatment
* Inability to understand or may not comply with test requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
unacceptable toxicity | 1 year
  "Unacceptable toxicity" is defined as any of the following toxicities: >1 episode of grade 3/4 neutropenia or thrombocytopenia <75,000/μL (despite prior dose reduction) during chemoradiation any toxicity that results in >2 week cumulative delay in chemoradiation any toxicity that is attributed to durvalumab which results in a delay of >8 weeks in surgery, i.e. surgery >16 weeks from the end of radiation, for a potentially operable patient any reason that is attributed to durvalumab which leads to death within 30 days of surgery
pathologic complete response rate, pCR | 1 year
major pahological response, MPR | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: chen ming, MD, Principal Investigator — Zhejiang Cancer Hospital; chen qixun, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shen D, Li R, She Y, Liu X, Huang Y, Ji Y, Chen K, Song Z, Chen R, Li X, Zhao Q, Chen Q, Chen M. PRDM1+ Malignant Cells Mediate an Immunosuppressive Landscape and Resistance to Neoadjuvant Chemoradiotherapy and Immunotherapy in Esophageal Squamous Cell Carcinoma. Adv Sci (Weinh). 2026 Jan 20:e15207. doi: 10.1002/advs.202515207. Online ahead of print. PMID 41556358